CLINICAL TRIAL: NCT00923273
Title: A Phase II Trial of Pemetrexed (Alimta [Registered Trademark]) Combined With Sirolimus (Rapamycin, Rapamune [Registered Trademark]) in Subjects With Relapsed or Refractory NSCLC
Brief Title: Sirolimus and Pemetrexed to Treat Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Premature closure - investigator left the National Institutes of Health.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Arun Rajan, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 080078; 08-C-0078; NCT00636532 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Results first posted 2013-10-23 (Estimated); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Pemetrexed; Sirolimus; Non-Small Cell Lung Cancer; Phase I/II; mTOR Inhibitor; NSCLC; Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Pemetrexed; Sirolimus; Vitamin B 12; Folic Acid; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Treatment level 1 - 3mg load (Experimental): Sirolimus 3mg load/1mg/day; Pemetrexed 375mg/m^2
  Interventions: Drug: FDG-PET; Drug: Pemetrexed; Drug: Sirolimus; Dietary Supplement: Vitamin B12; Dietary Supplement: Folic acid tablets; Drug: Dexamethasone tablets
- Treatment level 2 - 6 mg load (Experimental): Sirolimus 6mg load/2mg/day; Pemetrexed 375mg/m^2
  Interventions: Drug: FDG-PET; Drug: Pemetrexed; Drug: Sirolimus; Dietary Supplement: Vitamin B12; Dietary Supplement: Folic acid tablets; Drug: Dexamethasone tablets
- Treatment level 3 - 6mg load (Experimental): Sirolimus 6mg load/2mg/day; Pemetrexed 375mg/m^2
  Interventions: Drug: FDG-PET; Drug: Pemetrexed; Drug: Sirolimus; Dietary Supplement: Vitamin B12; Dietary Supplement: Folic acid tablets; Drug: Dexamethasone tablets
- Treatment level 4 - 10 mg load (Experimental): Sirolimus 10mg load/3mg/day; Pemetrexed 500mg/m^2
  Interventions: Drug: FDG-PET; Drug: Pemetrexed; Drug: Sirolimus; Dietary Supplement: Vitamin B12; Dietary Supplement: Folic acid tablets; Drug: Dexamethasone tablets
- Treatment level 5 - 15 mg load (Experimental): Sirolimus 15mg load/5mg/day; Pemetrexed 500mg/m^2
  Interventions: Drug: FDG-PET; Drug: Pemetrexed; Drug: Sirolimus; Dietary Supplement: Vitamin B12; Dietary Supplement: Folic acid tablets; Drug: Dexamethasone tablets

INTERVENTIONS:
Drug: FDG-PET — PET CT will be performed at baseline and after two cycles of treatment.
  Other Names: fluorodeoxyglucose positron emission tomography
Drug: Pemetrexed
Drug: Sirolimus
Dietary Supplement: Vitamin B12 — 1000 micrograms intramuscularly every 63 days administered the preceding first dose of pemetrexed
  Other Names: Cobalamin
Dietary Supplement: Folic acid tablets — 1 mg dose every 63 days administered during the week preceding first dose of pemetrexed and will be continued for 21 days following last dose of pemetrexed.
  Other Names: Folate
Drug: Dexamethasone tablets — 4 mg dose twice daily the day before, the day of, and the day after pemetrexed.
  Other Names: Decadron

SUMMARY:
Background:

The drug pemetrexed is used to treat non-small cell lung cancer (NSCLC) that does not respond to standard therapy or that has recurred after standard therapy; however, only 9 in 100 patients respond to pemetrexed.

Sirolimus is a drug that blocks a protein in cells called mammalian target of rapamycin (mTOR). In cancer cells, mTOR is active when it should not be, allowing the cells to grow uncontrollably. This protein is unusually active in many cases of NSCLC. By blocking the activity of mTOR, sirolimus may make the cancer cells more responsive to treatment with pemetrexed.

Objectives:

To determine if sirolimus in combination with pemetrexed is safe and well tolerated in patients with NSCLC.

To determine the highest safe dose of pemetrexed combined with sirolimus.

To look at the ability of sirolimus and pemetrexed to fight NSCLC.

To learn how the body eliminates sirolimus and pemetrexed.

Eligibility:

Patients 18 years of age and older with NSCLC whose disease does not respond to standard therapy or has recurred after treatment with standard therapy.

Design:

Biopsy before treatment starts, if the tumor is easy to reach by bronchoscopy or can be done by needle biopsy. This procedure is optional.

Drug treatment, as follows:

* Day 1: Intravenous (through a vein) infusions of pemetrexed. Small groups (3 to 6) of patients are given pemetrexed at a certain dose level. If the first group experiences no significant side effects, the next group receives a higher dose. This continues in succeeding groups for up to five dose levels until the maximum tolerated study dose (highest dose that patients can be given safely) is determined.
* To lessen the side effects of pemetrexed, patients also receive a Vitamin B12 injection every 21 days, folic acid tablets daily, and dexamethasone tablets twice a day the day before, the day of, and the day after pemetrexed infusions.
* Days 1-21: Sirolimus tablets by mouth.

Evaluations during the treatment period:

* History and physical examinations, blood and urine tests, electrocardiogram.
* Disease evaluation with computed tomography (CT), positron emission tomography (PET) or magnetic resonance scans (MRI) scans....

DETAILED DESCRIPTION:
Background:

* Lung cancer is the most deadly cancer due to late stage of diagnosis and intrinsic resistance to chemotherapy.
* Pemetrexed is a well tolerated Food and Drug Administration (FDA)-approved second line chemotherapeutic agent with a 9% response rate.
* Increasing the efficacy of pemetrexed could provide clinical benefit for patients with refractory NSCLC.
* Inhibition of the phosphoinositide 3-kinase (PI3K)/protein kinase B (Akt)/mTOR pathway may increase response to chemotherapy.
* Combining sirolimus, an mTOR inhibitor, with pemetrexed could improve patient outcomes.

Objectives:

* Determine the safety, tolerability, pharmacokinetics (PKs), and maximum tolerated dose (MTD) of the combination of sirolimus with pemetrexed in subjects with NSCLC subjects with activation of the Akt/mTOR pathway.
* Determine the clinical response rate at the MTD of sirolimus plus pemetrexed in NSCLC subjects.
* Determine effects of sirolimus on activation of the PI3K/Akt/mTOR pathway in peripheral blood mononuclear cells (PBMCs) and/or tumor tissues, to determine metabolic changes using PET scans, and measure PKs.

Eligibility:

- Adults with refractory or relapsed NSCLC regardless of mTOR pathway activation are permitted to enroll in the trial.

Design:

* Phase I followed by Phase II study
* For phase I/II subjects, documentation of mTOR pathway activation is not mandatory. If accessible, tissue will be obtained at baseline and following two cycles of therapy or at time of progression, whichever occurs first. Tumor tissue will be obtained at baseline and after two cycles of therapy or at time of progression, whichever occurs first. All subjects will have pathway analysis using PBMCs at baseline, day 8 and every two cycles of therapy or at time of progression, whichever occurs first. Cycle 1 is 28 days in length and all others 21 days.
* Each dose level incorporates a lead-in period of sirolimus alone that will allow for correlations of dose level, pharmacokinetics, and biologic effects.
* The phase I portion of the study has 5 dose cohorts beginning below the FDA approved doses for both agents. There are 3 dose escalations for sirolimus and 2 for pemetrexed. Up to 30 subjects may enroll in the phase I study.
* The Phase II portion will utilize the MTD from the Phase I and enroll up to 60 subjects.
* Sirolimus will be administered by mouth daily, and pemetrexed will be administered intravenously every 21 days until unacceptable toxicity or disease progression.
* Clinical imaging (CT or MRI) and a PET CT will be obtained at baseline and after two cycles of treatment. Clinical imaging will be performed every two cycles until disease progression.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Histologically documented non small cell lung cancer (NSCLC) that is confirmed by the Laboratory of Pathology at the Clinical Center/National Institutes of Health (NIH) or the Laboratory of Pathology at National Naval Medical Center (NNMC).
  2. Tumor biopsy will be requested from all study subjects unless the procedure poses too great a risk. If the subject declines, he or she may still participate in the study. We will ask subjects not undergoing biopsy to provide 6 unstained slides or a tissue block of archived tissue for immunohistochemistry (IHC) evaluation. Tumors from subjects enrolling in the phase II portion of the study will be analyzed retrospectively to demonstrate mammalian target of rapamycin (mTOR) activation as assessed by immunohistochemistry in a fresh biopsy. mTOR activation will be defined using distribution and intensity of staining for phosphorylation of mTOR, or its downstream substrates S6 kinase (S6K), and S6. Standard operating procedures (SOPs) describing the acquisition and handling of PBMCs and tissues are outlined in appendix 10.3 and 10.4. At a minimum, a total score (sum of intensity and distribution scores) of 2 for phospho-S6 or phospho-mTOR (S2448) mTOR will be required to determine that mTOR is active. Either measurement will be sufficient to ascertain that mTOR is active. Measurement of phosphorylation of Akt, factor 4E binding protein 1 (4E-BP1), and total levels of thymidylate synthase (TS) will also be measured, but are not part of the eligibility requirements. In the event of limited tissue availability, the stains will be prioritized as follows: S6, mTOR, S6K, Akt (S473), Akt (T308), and TS. Phosphorylation of S6 correlates most closely with mTOR activity, while phosphorylation of mTOR at S2448 best predicts response to sirolimus.
  3. Tissue from the time of original diagnosis will be adequate for enrollment on study. Optional fresh tissue biopsy must be obtained AFTER their most recent chemotherapy (including small molecule or targeted therapy) or radiation therapy. Tumors that can be biopsied percutaneously (with or without computed tomography (CT)/ultrasound guidance) or via bronchoscopy will be considered accessible if there are no other competing risk factors such as coagulopathy, hypoxemia, unstable cardiovascular disease, uncontrolled pain, or inability to give informed consent.
  4. Individuals with relapsed NSCLC who have received at least one standard chemotherapeutic regimen are eligible. Patients who received adjuvant chemotherapy and then relapse or recur less than or equal to 12 months after completion of chemotherapy will be eligible. Patients who received adjuvant chemotherapy and relapse greater than 12 months after completion of chemotherapy should receive frontline therapy for metastatic disease before enrollment, as should individuals who initially present with incurable disease that is chemotherapy naive. Individuals unwilling to receive standard front line therapy for metastatic lung cancer may enroll.
  5. Patients must have not received any chemotherapy, biological, or radiation therapy in the 21 days prior to protocol enrollment. All previous chemo and radiation therapy induced toxicities must have resolved to grade 1 or less prior to enrollment.
  6. Because sirolimus may affect the efficacy of hormonal birth control via cytochrome P450 3A4 (CYP 3A4), study subjects of child bearing potential must be willing to use barrier birth control while receiving sirolimus therapy and for 12 weeks after discontinuation of sirolimus.
  7. Patients must have measurable disease for the phase II portion of the study.
  8. Age greater than or equal to 18 years of age.
  9. Eastern Cooperative Oncology Group (ECOG) performance score of 0-2.
  10. An expected survival of at least 3 months.
  11. Patients must have the capacity to provide informed consent and demonstrate willingness to comply with an oral regimen.
  12. Patients must have normal organ and marrow function as defined below:
* Absolute neutrophil count greater than or equal to 1,500/mL.
* Platelets greater than or equal 100,000/mL.
* Total bilirubin less than 1.5 times upper limit of institutional normal.
* Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT) less than 2.5 times upper limit of institutional normal.
* Alanine aminotransferase (ALT) serum glutamic pyruvic transaminase (SGPT) less than 2.5 times upper limit of institutional normal.
* Creatinine Estimated creatinine clearance as calculated using the modification of diet in renal disease (MDRD) equation must be greater than or equal to 60ml/min/1.73m^2. The formula to be used is MDRD: 186 times (Scr)(-1.154) times (Age)(0.203) times (0.742 if female) times (1.212 if African American)
* Serum triglycerides less than or equal to 2.5 times upper limit of normal; serum cholesterol less than or equal 300 mg/dl (includes subjects with familial and acquired hyperlipidemia).

  13. Subjects on steroids must be on a stable or tapering dose of less than or equal 20 mg/day of prednisone (or equivalent dose of another glucocorticoid) for at least one week prior to study entry.

EXCLUSION CRITERIA:

1. Human immunodeficiency virus (HIV) positive patients.
2. Pregnant or lactating women.
3. Patients who received pemetrexed previously for Phase 1 only. Patients with prior pemetrexed are eligible for Phase 2.
4. Patients who have had prior therapy with mTOR inhibitors such as sirolimus or its analogues within six months.
5. Any concurrent therapy with chemotherapeutic agents or biologic agents or radiation therapy.
6. Subjects with brain metastases may participate if the metastases are asymptomatic. Subjects are ineligible if brain metastases are symptomatic.
7. Patients who are on the following drugs that modulate CYP3A4 and cannot replace these medications with other equivalent medications for the period of the study: amprenavir, atazanavir, bromocriptine, cimetidine, clarithromycin, clotrimazole, cyclosporine, danazol, diltiazem, erythromycin, fluconazole, fosamprenavir, other HIV protease inhibitors, indinavir, itraconazole, ketoconazole, metoclopramide, nefazodone, nelfinavir, nicardipine, nifedipine, ritonavir, saquinavir, telithromycin, troleandomycin (TAO), verapamil, voriconazole, nevirapine, rifampicin, rifampin, rifabutin, rifapentine, phenytoin, carbamazepine, phenobarbital, and St. John's Wort.
8. Subjects taking non steroidal anti-inflammatory agents who are unable to stop or replace the agents for the 5 days prior to and the 2 days after pemetrexed will not be eligible.
9. Patients who have received live vaccines in the past 21 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-02-29 (Actual); Primary Completion 2013-03-10 (Actual); Study Completion 2013-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arun Rajan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jemal A, Murray T, Ward E, Samuels A, Tiwari RC, Ghafoor A, Feuer EJ, Thun MJ. Cancer statistics, 2005. CA Cancer J Clin. 2005 Jan-Feb;55(1):10-30. doi: 10.3322/canjclin.55.1.10. PMID 15661684
- [Background] Schiller JH, Harrington D, Belani CP, Langer C, Sandler A, Krook J, Zhu J, Johnson DH; Eastern Cooperative Oncology Group. Comparison of four chemotherapy regimens for advanced non-small-cell lung cancer. N Engl J Med. 2002 Jan 10;346(2):92-8. doi: 10.1056/NEJMoa011954. PMID 11784875
- [Background] Fossella FV, DeVore R, Kerr RN, Crawford J, Natale RR, Dunphy F, Kalman L, Miller V, Lee JS, Moore M, Gandara D, Karp D, Vokes E, Kris M, Kim Y, Gamza F, Hammershaimb L. Randomized phase III trial of docetaxel versus vinorelbine or ifosfamide in patients with advanced non-small-cell lung cancer previously treated with platinum-containing chemotherapy regimens. The TAX 320 Non-Small Cell Lung Cancer Study Group. J Clin Oncol. 2000 Jun;18(12):2354-62. doi: 10.1200/JCO.2000.18.12.2354. PMID 10856094
- [Derived] Komiya T, Memmott RM, Blumenthal GM, Bernstein W, Ballas MS, De Chowdhury R, Chun G, Peer CJ, Figg WD, Liewehr DJ, Steinberg SM, Giaccone G, Szabo E, Kawabata S, Tsurutani J, Rajan A, Dennis PA. A phase I/II study of pemetrexed with sirolimus in advanced, previously treated non-small cell lung cancer. Transl Lung Cancer Res. 2019 Jun;8(3):247-257. doi: 10.21037/tlcr.2019.04.19. PMID 31367538
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2008-C-0078.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: DL5 wasn't tolerated. We expanded DL4, had 1 DLT of gr. 3 infection that was possibly related to study drugs or his cancer and declining health. The last subject on DL4 had gr. 4 neutropenia that lasted <7days. We believe this wasn't significant and a lack of foresight to add length of neutropenia as DLT. IRB allowed DL4 with DLT stopping rule.
Groups:
- Treatment Level 1: 3mg Load: Sirolimus 3mg load/1mg/day; Pemetrexed 375mg/m^2
- Treatment Level 2: 6mg Load: Sirolimus 6mg load/2mg/day; Pemetrexed 375mg/m^2
- Treatment Level 3: 6mg Load: Sirolimus 6mg load/2mg/day; Pemetrexed 500mg/m^2
- Treatment Level 4: 10mg Load: Sirolimus 10mg load/3mg/day; Pemetrexed 500mg/m^2
- Treatment Level 5: 15mg Load: Sirolimus 15mg load/5mg/day; Pemetrexed 500mg/m^2
Period: Phase I Treatment Period
Arm/Group | Treatment Level 1: 3mg Load | Treatment Level 2: 6mg Load | Treatment Level 3: 6mg Load | Treatment Level 4: 10mg Load | Treatment Level 5: 15mg Load
Started | 4 (The phase I portion will establish the maximum tolerated dose. 4 subjects peme naive.) | 3 (3 subjects peme naive.) | 3 (3 subjects peme naive.) | 7 (3 subjects initially enrolled and 4 subjects added after dose level 5; peme naive.) | 5 (5 subjects peme naive.)
Completed | 4 | 3 | 3 | 7 | 5
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Phase II Treatment Period
Arm/Group | Treatment Level 1: 3mg Load | Treatment Level 2: 6mg Load | Treatment Level 3: 6mg Load | Treatment Level 4: 10mg Load | Treatment Level 5: 15mg Load
Started | 0 (The phase II portion will utilize the MTD from the phase I portion.) | 0 | 0 | 27 (Includes 8 subjects with prior peme;12 subjects who were peme naive; 7 subjects rolled over from phI) | 0
Completed | 0 | 0 | 0 | 20 | 0
Not Completed | 0 | 0 | 0 | 7 | 0
Not completed — NE-brain mets/met disease prior enrollmt | 0 | 0 | 0 | 1 | 0
Not completed — NE-not complete 2Cy trmt/no imaging done | 0 | 0 | 0 | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Level 4: 10 mg Load: Sirolimus 10mg load/3mg/day; Pemetrexed 500mg/m^2
- Total: Total of all reporting groups
Arm/Group | Treatment Level 1: 3mg Load | Treatment Level 2: 6mg Load | Treatment Level 3: 6mg Load | Treatment Level 4: 10 mg Load | Treatment Level 5: 15mg Load | Total
Number analyzed (Participants) | 4 | 3 | 3 | 27 | 5 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 1 | 18 | 4 | 25
  >=65 years | 2 | 3 | 2 | 9 | 1 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.65 (7.84) | 71.57 (3.76) | 61.7 (24.74) | 59.5 (11.48) | 56.08 (10.75) | 60.6 (11.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 14 | 2 | 21
  Male | 2 | 1 | 2 | 13 | 3 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2 | 0 | 4
  Not Hispanic or Latino | 4 | 2 | 2 | 25 | 5 | 38
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 4 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 4 | 0 | 6
  White | 4 | 0 | 1 | 18 | 5 | 28
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 3 | 3 | 27 | 5 | 42

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD) of Pemetrexed
Description: The phase I component of the study are to determine the safety and tolerability of pemetrexed in human subjects with non small cell lung cancer (NSCLC), and to determine the maximum tolerated dose.
Time Frame: 5 weeks
Measure: Number; unit: mg/m^2
Groups:
- Treatment Level 1: 3mg Load: Sirolimus 3mg load/1mg/day; Pemetrexed 375mg/m^2 All subjects completed the intervention and phase I outcome measure.
- Treatment Level 2: 6mg Load: Sirolimus 6mg load/2mg/day; Pemetrexed 375mg/m^2 All subjects completed the intervention and phase I outcome measure.
- Treatment Level 3: 6mg Load: Sirolimus 6mg load/2mg/day; Pemetrexed 500mg/m^2 All subjects completed the intervention and phase I outcome measure.
- Treatment Level 4: 10mg Load: Sirolimus 10mg load/3mg/day; Pemetrexed 500mg/m^2 All subjects completed the intervention and phase I outcome measure.
- Treatment Level 5: 15mg Load: Sirolimus 15mg load/5mg/day; Pemetrexed 500mg/m^2 All subjects completed the intervention and phase I outcome measure.
Arm/Group | Treatment Level 1: 3mg Load | Treatment Level 2: 6mg Load | Treatment Level 3: 6mg Load | Treatment Level 4: 10mg Load | Treatment Level 5: 15mg Load
Number analyzed (Participants) | 4 | 3 | 3 | 7 | 5
mg/m^2 | 500 | 500 | 500 | 500 | 500

2. Secondary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v3.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 45 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Level 1: 3mg Load | Treatment Level 2: 6mg Load | Treatment Level 3: 6mg Load | Treatment Level 4: 10 mg Load | Treatment Level 5: 15mg Load
Number analyzed (Participants) | 4 | 3 | 3 | 27 | 5
Participants
  Subjects from phase I | 4 | 3 | 3 | 7 | 5
  8subjects prior peme & 12 subjects peme naive | 0 | 0 | 0 | 20 | 0

3. Primary Outcome: Phase II: Clinical Response Rate
Description: Clinical response is assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response (CR) is disappearance of all target lesions. Partial response (PR) at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started. Progressive disease (PD) is at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: 21 weeks
Population: By formal criteria in the protocol, DL4 exceeds the MTD, and DL 3 would be expanded by 3 subjects to confirm it's tolerability. We believe that DL4 is safe, and that the observed DLTs at this DL are related to enrollment of a subject with a borderline performance status, and the omission of defining length of neutropenia as a DLT.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Level 4: 10mg Load: Sirolimus 10mg load/3mg/day; Pemetrexed 500mg/m^2
  Includes 8 subjects with prior peme; 12 subjects who were peme naive;and 7 subjects rolled over from ph I
Arm/Group | Treatment Level 4: 10mg Load
Number analyzed (Participants) | 27
Participants
  Complete response | 0
  Partial response | 5
  Stable disease | 13
  Progressive disease | 2
  Not evaluable | 7

4. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD) of Sirolimus
Description: The phase I component of the study are to determine the safety and tolerability of sirolimus in human subjects with non small cell lung cancer (NSCLC), and to determine the maximum tolerated dose.
Time Frame: 5 weeks
Measure: Number; unit: mg/m^2
Arm/Group | Treatment Level 1: 3mg Load | Treatment Level 2: 6mg Load | Treatment Level 3: 6mg Load | Treatment Level 4: 10mg Load | Treatment Level 5: 15mg Load
Number analyzed (Participants) | 4 | 3 | 3 | 7 | 5
mg/m^2 | 10 | 10 | 10 | 10 | 10

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 45 months.
Arm/Group | Treatment Level 1: 3mg Load | Treatment Level 2: 6mg Load | Treatment Level 3: 6mg Load | Treatment Level 4: 10 mg Load | Treatment Level 5: 15mg Load
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 1/3 | 0/27 | 0/5
Serious Adverse Events (participants affected / at risk) | 2/4 | 1/3 | 0/3 | 7/27 | 1/5
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 3/3 | 27/27 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Level 1: 3mg Load (N=4) | Treatment Level 2: 6mg Load (N=3) | Treatment Level 3: 6mg Load (N=3) | Treatment Level 4: 10 mg Load (N=27) | Treatment Level 5: 15mg Load (N=5)
Edema: limb (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Death not associated with CTCAE term: Disease progression NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — (fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0x10e9/L): lung (pneumonia)
Infection with normal ANC or Grade 1 or 2 neutrophils: lung (pneumonia) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pulmonary/Upper respiratory - Other (specify, pulmonary infiltrate, right lung) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CD4 count (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholesterol, serum-high (hypercholesteremia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Creatinine (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Level 1: 3mg Load (N=4) | Treatment Level 2: 6mg Load (N=3) | Treatment Level 3: 6mg Load (N=3) | Treatment Level 4: 10 mg Load (N=27) | Treatment Level 5: 15mg Load (N=5)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 1 (7) | 2 (4) | 1 (1) | 6 (20) | 3 (13)
AST/SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 3 (9) | 2 (2) | 0 (0) | 5 (11) | 3 (10)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2 (11) | 3 (14) | 3 (8) | 7 (16) | 5 (13)
Alkaline phosphatase (Metabolism and nutrition disorders) | 4 (7) | 2 (3) | 1 (2) | 3 (6) | 2 (5)
Anorexia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 16 (19) | 4 (7)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 2 (5) | 1 (1) | 1 (2) | 3 (16) | 1 (1)
Cholesterol, serum-high (hypercholesteremia) (Metabolism and nutrition disorders) | 1 (2) | 2 (3) | 1 (2) | 4 (10) | 2 (2)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 6 (6) | 2 (3)
Creatinine (Metabolism and nutrition disorders) | 1 (8) | 1 (1) | 1 (1) | 3 (5) | 3 (12)
Diarrhea (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0) | 13 (15) | 2 (2)
Distention/bloating, abdominal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dry eye syndrome (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 7 (10) | 3 (5)
Edema: limb (Blood and lymphatic system disorders) | 1 (4) | 1 (1) | 0 (0) | 4 (4) | 2 (3)
Edema: trunk/genital (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FEV(1) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 (3) | 1 (1) | 0 (0) | 18 (27) | 5 (13)
Fever (General disorders) | 2 (2) | 1 (1) | 1 (1) | 8 (9) | 1 (1) — (in the absence of neutropenia, where neutropenia is defined as ANC <1.0x10e9/L)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
GGT (gamma-Glutamyl transpeptidase) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal - Other (Specify, bloating) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glomerular filtration rate (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (16) | 2 (2) | 1 (1) | 9 (32) | 4 (14)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hemoglobin (Metabolism and nutrition disorders) | 3 (23) | 3 (17) | 3 (6) | 12 (26) | 5 (34)
Hemorrhage/Bleeding - Other (Specify, nose) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection - Other (Specify, pneumonia) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (General disorders) | 3 (4) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (7) | 2 (4) | 3 (5) | 9 (23) | 2 (8)
Lymphopenia (Blood and lymphatic system disorders) | 3 (14) | 2 (15) | 3 (3) | 17 (49) | 5 (29)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 2 (3) | 1 (5) | 0 (0) | 5 (10) | 2 (2)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 2 (8) | 1 (3) | 1 (2) | 11 (22) | 4 (10)
Mood alteration: anxiety (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Mood alteration: depression (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Mucositis/stomatitis (clinical exam): oral cavity (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 6 (9) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 14 (16) | 4 (5)
Neuropathy: sensory (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (4) | 2 (2) | 2 (4) | 10 (20) | 2 (7)
PTT (Partial thromboplastin time) (Blood and lymphatic system disorders) | 2 (6) | 1 (2) | 3 (11) | 3 (7) | 4 (7)
Pain - Other (Specify, L rib; R costal margin; shoulder) (General disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain: Abdomen NOS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 6 (8) | 0 (0)
Pain: Bone (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain: extremity-limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain: oral cavity (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 2 (14) | 2 (5) | 1 (2) | 13 (36) | 3 (7)
Platelets (Blood and lymphatic system disorders) | 1 (7) | 2 (5) | 3 (4) | 9 (17) | 4 (9)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 2 (2)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (4) | 1 (5) | 0 (0) | 2 (4) | 2 (3)
Proteinuria (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Pruritis/itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Rash/acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 11 (12) | 2 (2)
Renal/Genitourinary - Other (Specify, renal insufficiency) (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rigors/chills (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 4 (6) | 2 (13) | 1 (2) | 11 (32) | 4 (11)
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Speech impairment (e.g., dysphagia or aphasia) (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular and nodal arrhythmia: sinus tachycardia (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 4 (4) | 1 (1)
Sweating (diaphoresis) (General disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 1 (4) | 2 (2) | 1 (1) | 2 (4) | 1 (1)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vital capacity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (3) | 1 (1) | 9 (13) | 3 (6)
Watery eye (epiphora, tearing) (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Ocular surface disease (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain: back (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Pain: eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain: head/headache (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 6 (6) | 2 (2)
Pain: rectum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 1 (1)
CNS cerebrovascular ischemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain: joint (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Ascites (non-malignant) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Auditory/Ear - Other (Specify, hearing loss right side) (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CD4 count (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 15 (37) | 3 (4)
Cardiac troponin I (cTnl) (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatology/Skin - Other (Specify, decubitus) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0)
INR (International Normalized Ratio of prothrombin time) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — (ANC<1.0x10e9/L): oral cavity-gum (gingivitis)
Infection - Other (Specify, URI) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils: bladder (urinary) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils: oral cavity-gums (gingivitis) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils: sinus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils: skin (cellulitis) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 1 (1)
Mucositis/stomatitis (functional/symptomatic): oral cavity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Muscle weakness, genralized or specific area (not due to neuropathy): extraocular (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness, genralized or specific area (not due to neuropathy): extremity-lower (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Muscle weakness, genralized or specific area (not due to neuropathy): whole body/generalized (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nail changes (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain: Other (Specify) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) — chest pleuritic; left thigh; right rib; right shin; due to fall-hip
Pain: dental/teeth/periodontal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain: neuralgia/peripheral nerve (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain: pelvis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pain: throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 2 (2)
Personality/behavioral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash: erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Supraventricular and nodal arrhythmia: atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision-blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Voice changes/dysarthia (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Weight gain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight loss (General disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (10) | 0 (0)
Gastrointestinal - Other (Specify, early satiety) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary/Upper respiratory - Other (Specify, mild drain. from podt throat) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain: Anus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain: Stomach (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 3 (3) | 0 (0)
Infection (documented clinically or microbiologically) with Grade 3 or 4 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — neutrophils (ANC <1.0x10e9/L): urinary tract NOS
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Cardiac arrhythmia (Other (Specify, tavhycardia) (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Edema: head and neck (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Flushing (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Febrile neutropenia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — (fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0x10e9/L, fever >=38.5 degrees C)
Heartburn/dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (8) | 1 (1)
Hemorrhage, pulmonary/upper respiratory:bronchopulmonary NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 2 (3)
Mood alteration:agitation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pain: chest wall (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (8) | 1 (1)
Pain: chest/thorax NOS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain: muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 1 (1)
Ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary frequency/urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pulmonary/Upper respiratory - Other (Specify, pulmonary infiltrates) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Auditory/Ear - Other (Specify, congestion R/ear) (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain - Other (Specify, left elbow; left flank; left trunk) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Renal/Genitourinary - Other (Specify, ARI) (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage, pulmonary/upper respiratory: nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Urine color change (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hemorrhage, pulmonary/upper respiratory: Bronchus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils: Lung (pneumonia) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils: Rectum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with unknown ANC: Lung (pneumonia) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with unknown ANC: Skin (cellulitis) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with unknown ANC: upper airway NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obstruction/stenosis of airway: Bronchus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2012-11-16): https://cdn.clinicaltrials.gov/large-docs/73/NCT00923273/Prot_SAP_000.pdf
  • Informed Consent Form (2012-03-27): https://cdn.clinicaltrials.gov/large-docs/73/NCT00923273/ICF_001.pdf